CLINICAL TRIAL: NCT01981980
Title: Comparison of the Effects of Carboxytherapy and Radiofrequency on Skin Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adriana Clemente Mendonça (Other)
Responsible Party: Sponsor-Investigator, Adriana Clemente Mendonça, Professor, Universidade Federal do Triangulo Mineiro
Organization: Universidade Federal do Triangulo Mineiro (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CEP1362
Record Dates: First submitted 2013-10-29; First posted 2013-11-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Skin Aging; Skin Rejuvenation
Keywords: Carbon dioxide; Carboxytherapy; Radiofrequency
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carboxytherapy (Experimental): It was administered using the beveled end of a 30G ½ needle introduced in the skin in an angle of approximately 30ºC and delivered at a velocity of 40 mL/min. The total quantity of CO2 infused was approximately 20 mL (0,3 to 0,6 mL/kg of patient's body weight) encompassing the whole delimited area.
  Interventions: Other: Carboxytherapy
- Radiofrequency (Experimental): The epidermal temperature was controlled using an infrared thermometer monitored to reach 40ºC and treatment time was of five minutes starting after having reached this temperature.
  Interventions: Other: Radiofrequency

INTERVENTIONS:
Other: Carboxytherapy — Carboxytherapy was performed on the right side and RF on the left side. CA was administered using the beveled end of a 30G ½ needle introduced in the skin in an angle of approximately 30ºC and delivered at a velocity of 40 mL/min. The total quantity of CO2 infused was approximately 20 mL (0,3 to 0,6 mL/kg of patient's body weight) encompassing the whole delimited area.
  Other Names: Physical Therapy treatment
  Arms: Carboxytherapy
Other: Radiofrequency — The epidermal temperature was controlled using an infrared thermometer monitored to reach 40ºC and treatment time was of five minutes starting after having reached this temperature.
  Arms: Radiofrequency

SUMMARY:
Carboxytherapy (CA) refers to the cutaneous and subcutaneous administration of carbon dioxide gas [CO2] for therapeutic purposes. Radiofrequency (RF) is a method that uses electric current to generate heat into the layers of the skin and the subcutaneous tissue. Both techniques are indicated to the treatment of skin laxity. The aim of this study was to compare the effects of CA an RF on human skin. Methods: Eight patients who underwent abdominoplasty surgery received a single procedure of both treatments. Untreated skin was used as control. In an area of 49 cm2 (7 x 7 cm) in the infra-umbilical region CA was performed on the right and RF on the left side. Sample collection period ranged from zero to 120 days. CA was administered at a velocity of 40 ml/min, and the total quantity of CO2 infused was approximately 20ml. RF was carried out in a temperature higher than 40ºC on the epidermis for 5 minutes after reaching this temperature.

DETAILED DESCRIPTION:
Untreated skin was used as control. In an area of 49 cm2 (7 x 7 cm) in the infra-umbilical region CA was performed on the right side and RF on the left side. CA was administered using the beveled end of a 30G ½ needle introduced in the skin in an angle of approximately 30ºC and delivered at a velocity of 40 mL/min. The total quantity of CO2 infused was approximately 20 mL (0,3 to 0,6 mL/kg of patient's body weight) encompassing the whole delimited are. For the RF treatment, the epidermal temperature was controlled using an infrared thermometer monitored to reach 40ºC and treatment time was of five minutes starting after having reached this temperature. Sample collection varied from zero to 120 days after application. The samples were then fixed, cut in paraffin (5 µm) and stained with Picro sirus and Weigert. Morphological analyses were acquired using a Zeiss Axiophot® microscope, and they were processed using Adobe Photoshop®.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent abdominoplasty surgery and agree to participate to this study

Exclusion Criteria:

* patients been treated with corticosteroids or anti-inflammatory during the period of the protocol, with cancer or other change that contraindicated the application of carboxytherapy and radiofrequency

Ages: 27 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Effect on Skin morphology treatment with Carboxytherapy and Radiofrequency at the same day of a single session | same 1 day of a single session treatment
  Evaluation of elastic fiber and collagen remodeling from skin treated or not with Carboxytherapy and Radiofrequency. Samples were obtained from one patient who underwent abdominoplasty surgery. The samples were fixed, processed to paraffin and stained with Picro sirus and Weigert. Images were acquired using a Zeiss Axiophot® microscope, and they were processed using Adobe Photoshop®.

SECONDARY OUTCOMES:
Effect on Skin morphology treatment with Carboxytherapy and Radiofrequency at the forth day after a single session | 4th day after a single session
  Evaluation of elastic fiber and collagen remodeling from skin treated or not with Carboxytherapy and Radiofrequency. Samples were obtained from one patient who underwent abdominoplasty surgery. The samples were fixed, processed to paraffin and stained with Picro sirus and Weigert. Images were acquired using a Zeiss Axiophot® microscope, and they were processed using Adobe Photoshop®.

OTHER OUTCOMES:
Effect on Skin morphology treatment with Carboxytherapy and Radiofrequency at the 20th day after a single session | 20th day after a single session
  Evaluation of elastic fiber and collagen remodeling from skin treated or not with Carboxytherapy and Radiofrequency. Samples were obtained from one patient who underwent abdominoplasty surgery. The samples were fixed, processed to paraffin and stained with Picro sirus and Weigert. Images were acquired using a Zeiss Axiophot® microscope, and they were processed using Adobe Photoshop®.
Effect on Skin morphology treatment with Carboxytherapy and Radiofrequency at the 28th day after a single session | 28th day after a single
  Evaluation of elastic fiber and collagen remodeling from skin treated or not with Carboxytherapy and Radiofrequency. Samples were obtained from one patient who underwent abdominoplasty surgery. The samples were fixed, processed to paraffin and stained with Picro sirus and Weigert. Images were acquired using a Zeiss Axiophot® microscope, and they were processed using Adobe Photoshop®.
Effect on Skin morphology treatment with Carboxytherapy and Radiofrequency at the 44th day after a single session | 44th day after a single session
  Evaluation of elastic fiber and collagen remodeling from skin treated or not with Carboxytherapy and Radiofrequency. Samples were obtained from one patient who underwent abdominoplasty surgery. The samples were fixed, processed to paraffin and stained with Picro sirus and Weigert. Images were acquired using a Zeiss Axiophot® microscope, and they were processed using Adobe Photoshop®.
Effect on Skin morphology treatment with Carboxytherapy and Radiofrequency at the 61th day after a single session | 61th day after a single session
  Evaluation of elastic fiber and collagen remodeling from skin treated or not with Carboxytherapy and Radiofrequency. Samples were obtained from one patient who underwent abdominoplasty surgery. The samples were fixed, processed to paraffin and stained with Picro sirus and Weigert. Images were acquired using a Zeiss Axiophot® microscope, and they were processed using Adobe Photoshop®.
Effect on Skin morphology treatment with Carboxytherapy and Radiofrequency at the 117th day after a single session | 117th day after a single session
  Evaluation of elastic fiber and collagen remodeling from skin treated or not with Carboxytherapy and Radiofrequency. Samples were obtained from one patient who underwent abdominoplasty surgery. The samples were fixed, processed to paraffin and stained with Picro sirus and Weigert. Images were acquired using a Zeiss Axiophot® microscope, and they were processed using Adobe Photoshop®.
Effect on Skin morphology treatment with Carboxytherapy and Radiofrequency at the 120th day after a single session | 120th day after a single session
  Evaluation of elastic fiber and collagen remodeling from skin treated or not with Carboxytherapy and Radiofrequency. Samples were obtained from one patient who underwent abdominoplasty surgery. The samples were fixed, processed to paraffin and stained with Picro sirus and Weigert. Images were acquired using a Zeiss Axiophot® microscope, and they were processed using Adobe Photoshop®.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana C Mendonça, Ph.D., Principal Investigator — Federal University of Triângulo Mineiro
Locations (1):
- Adriana Clemente Mendonça, Uberaba, Minas Gerais, Brazil